CLINICAL TRIAL: NCT07064863
Title: BCG-TIME: Improving Response to Bacillus Calmette Guerin Immunotherapy in High-risk Non-muscle Invasive Bladder Cancer Via a Tumor Immune MicroEnvironment Based Biomarker.
Brief Title: A Tumor Immune Biomarker Guided Approach for Improving Response to BCG in Patients With High-risk NMIBC.
Acronym: BCG-TIME
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Queen's University, Kingston, Ontario (Other)
Responsible Party: Principal Investigator, Madhuri Koti, Associate Professor, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6043613
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: NMIBC; Non-Muscle Invasive Bladder Urothelial Carcinoma; Bladder (Urothelial, Transitional Cell) Cancer; Urothelial Carcinoma Bladder
Keywords: BCG; NMIBC; Gemcitabine; Tumor Immune MicroEnvironment; Systemic immunity; Mucosal immune response; Immune Biomarker
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Neoplasms | interventions — Gemcitabine; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravesical Gemcitabine + BCG (Experimental): Patients will be recruited to treatment with gemcitabine at week 0 following which BCG (50 mg, TICE strain) will be administered once every week for a total of 5 instillations.
  Interventions: Drug: Gemcitabine + BCG
- Intravesical Bacillus Calmette-Guérin (BCG) (Active Comparator): 6 intravesical instillations of BCG (50 mg, TICE strain) at weekly intervals.
  Interventions: Drug: BCG (TICE strain)

INTERVENTIONS:
Drug: Gemcitabine + BCG — Patients will receive a single intravesical instillation of gemcitabine (2000 mg) at week 0 followed by weekly BCG (50 mg of TICE strain) for a total of 5 instillations. Biopsy will be conducted within three months of completing the induction phase.
  Arms: Intravesical Gemcitabine + BCG
Drug: BCG (TICE strain) — Patients will receive intravesical BCG (50 mg, TICE strain) at weekly intervals for a total of 6 instillations. Biopsy will be performed within 3 months of completing the induction phase.
  Arms: Intravesical Bacillus Calmette-Guérin (BCG)

SUMMARY:
This study is being conducted to establish a novel tumor tissue- and blood-based biomarker test to assess early systemic and local response to immunomodulation by BCG immunotherapy in patients with high-risk non-muscle invasive bladder cancer. Responses will be compared between patients with high-risk NMIBC who are being treated with standard of care BCG therapy and those treated with combination chemotherapy. Local and systemic immune monitoring assays will allow early identification of patients who will not benefit from BCG immunotherapy.

DETAILED DESCRIPTION:
BCG immunotherapy is the current gold standard for NMIBC. However, ~50% of patients will eventually experience recurrence or progression. Pre-treatment immune competence of the patient, the bladder microenvironment and systemic immune responses to immunomodulation by BCG govern effectiveness. The investigators intend to utilize a novel tumor tissue and blood based biomarker test to assess early systemic responses to standard of care BCG based immunotherapy as well as alternate strategies to enhance immune responses as measured systemically as well as based on early response rates (3 month complete response or 3 month recurrence). The goal of this study is to develop strategies to identify novel more effective anti-tumor immune responses for NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an initial diagnosis of NMIBC without previous exposure to BCG immunotherapy (BCG-naive).
* Patients with pathologic diagnosis of Ta or T1 high grade NMIBC with or without CIS.
* Participants older than 65 years of age.

Exclusion Criteria:

* Patients with prior exposure to BCG immunotherapy.
* Immunosuppressed patients on steroids, transplants etc.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
BCG ImmunoScore | 3 months
  Complete response at 3 months with no evidence of tumor recurrence as assessed by biopsy. Demonstrable immunological responses measured at weeks 2, and 5 post-treatment, based on a novel tissue and blood based immune biomarker.

SECONDARY OUTCOMES:
Recurrence free survival | 12 months
  Recurrence free survival at 12 months post treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No